CLINICAL TRIAL: NCT00742508
Title: A Study to Evaluate the Safety and Tolerability of SK&F-105517-D in Patients With Chronic Heart Failure- An Open-label Study to Evaluate the Safety and Tolerability, Pharmacokinetics and Pharmacodynamics of SK&F-105517-D in Patients With Chronic Heart Failure (Phase I/II Study)
Brief Title: A Phase I/II Clinical Study of SK&F-105517-D in Japanese Patients With Chronic Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRV110734
Record Dates: First submitted 2008-08-26; First posted 2008-08-27 (Estimated); Results first posted 2010-08-19 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-06

CONDITIONS: Heart Failure, Congestive
Keywords: carvedilol phosphate; ß-blocker; SK&F-105517-D; Chronic heart failure(CHF)
MeSH Terms: conditions — Heart Failure | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SK&F-105517-D group (Experimental): SK&F-105517-D 10-80 mg/day
  Interventions: Drug: SK&F-105517-D 10 mg capsule; Drug: SK&F-105517-D 20 mg capsule; Drug: SK&F-105517-D 40 mg capsule
- Carvedilol-IR group (Other): Carvedilol-IR 5-20 mg/day
  Interventions: Drug: Carvedilol-immediate release (IR) 2.5 mg tablet; Drug: Carvedilol-IR 10 mg tablet

INTERVENTIONS:
Drug: SK&F-105517-D 10 mg capsule — 1 capsule once a day
  Other Names: carvedilol phosphate
  Arms: SK&F-105517-D group
Drug: Carvedilol-immediate release (IR) 2.5 mg tablet — 1 or 2 tablet(s) twice a day
  Arms: Carvedilol-IR group
Drug: SK&F-105517-D 20 mg capsule — 1 capsule once a day
  Other Names: carvedilol phosphate
  Arms: SK&F-105517-D group
Drug: SK&F-105517-D 40 mg capsule — 1 or 2 capsule(s) once a day
  Other Names: carvedilol phosphate
  Arms: SK&F-105517-D group
Drug: Carvedilol-IR 10 mg tablet — 1 tablet twice a day
  Arms: Carvedilol-IR group

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of SK&F-105517-D in japanese patients with chronic heart failure.

ELIGIBILITY:
Inclusion criteria:

* Patients with symptomatically stable chronic heart failure (CHF) based on ischemic heart disease or dilated cardiomyopathy
* Patients who are maintained on basic heart failure therapy with angiotensin converting enzyme (ACE) inhibitors or angiotensin II receptor blocker (ARB) and their dosage/administration is not changed within 2 weeks
* Patients diagnosed with New York Heart Association (NYHA) class I to III
* Patients with a left ventricular ejection fraction (LVEF) between 25% and 45%

Exclusion Criteria:

* Patients contraindicated for ß-blockers
* Patients with occurrence of acute myocardial infarction within 2 weeks
* Patients with unstable angina, coronary spastic angina, or angina at rest
* Patients who have collected blood >400 mL within 4 months prior to screening or >200 mL within 1 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2008-08-28 (Actual); Primary Completion 2009-08-21 (Actual); Study Completion 2009-08-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (15):
- Japan (15):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Mie
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Ōita
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Wakayama

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kitakaze M, Sarai N, Ando H, Sakamoto T, Nakajima H. Safety and tolerability of once-daily controlled-release carvedilol 10-80 mg in Japanese patients with chronic heart failure. Circ J. 2012;76(3):668-74. doi: 10.1253/circj.cj-11-0210. Epub 2012 Jan 12. PMID 22240593
- See also: Results for study 110734 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/CRV110734?search=study&study_ids=110734#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: CRV110734 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: CRV110734 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: CRV110734 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: CRV110734 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: CRV110734 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants randomized to receive SK&F-105517-D underwent 2 weeks of observation, 8 weeks of Primary Evaluation, 4 weeks of Exploratory Evaluation, 2 weeks of dose-tapering, and 1 week of Follow-up period. Participants randomized to receive CRV-IR underwent 2 weeks of observation, 8 weeks of Primary Evaluation, and 1 week of Follow-up.
Groups:
- CRV-IR: In the 8-week Primary Evaluation Period (including the 2-week Run-in Period [from Week 0 as Baseline]), participants received an initial dose of an immediate-release (IR) formulation of carvedilol (CRV) as a 1.25 milligram (mg) tablet twice daily (BID) (2.5 mg/day) at Week 0, followed by an increased dose of CRV-IR 2.5 mg tablet BID (5 mg/day) at Week 1. The dose was then increased to 5 mg BID (10 mg/day) at Week 4, and finally to 10 mg BID (20 mg/day) at Week 6. The participants on CRV-IR were switched to the marketed CRV-IR in Week 1 of the Follow-up Period; the investigator or subinvestigator determined the dose of the marketed CRV-IR based on the last dose administered during the Primary Evaluation Period after confirming the safety and tolerability of the dose.
- SK&F-105517-D: In the 8-week Primary Evaluation Period (including the 2-week Run-in Period [from Week 0 as Baseline]), participants received a CRV-IR 1.25 mg and 2.5 mg tablet BID at Weeks 0 and 1, respectively. They then received a 10 mg extended-release capsule of carvedilol (SK&F-105517-D) once daily (OD) at Week 2; the dose was then increased to 20 mg OD and finally to 40 mg OD at 2-week intervals. The dose was increased from 40 mg to 60 mg and finally to 80 mg at 2-week intervals in the 4-week Exploratory Evaluation Period after confirming that each dose was well tolerated without safety concern and that the participant met all of the dose-escalation criteria. During the 2-week Dose-tapering Period set up to prepare for switch to the marketed CRV-IR, the dose of SK&F-105517-D was reduced to 60 mg OD and then to 40 mg OD at weekly intervals; SK&F-105517-D was then switched to the marketed CRV-IR 10 mg tablet BID in the 1-week Follow-up Period.
Period: 8-Week Primary Evaluation Period
Arm/Group | CRV-IR | SK&F-105517-D
Started | 22 | 19
Completed | 11 | 8
Not Completed | 11 | 11
Not completed — Adverse Event | 2 | 4
Not completed — Protocol Violation | 1 | 0
Not completed — Met Protocol-defined Stopping Criteria | 8 | 5
Not completed — Withdrawal by Subject | 0 | 2
Period: 4-Week Exploratory Evaluation Period
Arm/Group | CRV-IR | SK&F-105517-D
Started | 0 | 8
Completed | 0 | 7
Not Completed | 0 | 1
Not completed — Met Protocol-defined Stopping Criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CRV-IR | SK&F-105517-D | Total
Number analyzed (Participants) | 22 | 19 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.17) | 66.7 (12.00) | 64.6 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 20 | 18 | 38
Race/Ethnicity, Customized [Number; unit: participants]
  Asian-Japanese Heritage | 22 | 19 | 41

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events by Severity From Week 0 Through Week 8 (CRV-IR) or Week 14 (SK&F-105517-D)
Description: Drug-related adverse events (AEs) were defined as AEs that were judged to have a relationship with the investigational product by the investigator (or subinvestigator) with the use of clinical judgment and the Clinical Investigator Brochure to determine the relationship. Refer to adverse event information for type and frequency of adverse events.
Time Frame: Treatment Period from Week 0 (Baseline) to Week 8 and 1-week Follow-up Period (Week 9) for CRV-IR; Treatment Period from Week 0 (Baseline) to Week 14 and 1-week Follow-up Period (Week 15) for SK&F-105517-D
Population: Safety Population: all participants who received at least one dose of the investigational product
Measure: Number; unit: participants
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
participants
  Severe | 0 | 1
  Moderate | 2 | 5
  Mild | 9 | 10
  Severe (drug-related) | 0 | 1
  Moderate (drug-related) | 2 | 3
  Mild (drug-related) | 3 | 4

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) and Trough Plasma Concentration (Cmin) of S-carvedilol, R-carvedilol, and M4 Active Metabolite (SB-203231) at Week 8
Description: Maximum Plasma Concentration (Cmax) and Trough Plasma Concentration (Cmin) of S-carvedilol, R-carvedilol, and M4 active Metabolite (SB-203231) were measured. Participants in each treatment group were divided into 3 groups by pharmacokinetic sampling timing: Groups A, B, and C in the SK&F-105517-D group and Groups D, E, and F in the CRV-IR group. The analysis was performed on log-transformed data. Carvedilol is a racemic mixture. Non-selective β-blocking activity is shown by S-carvedilol, while α1-blocking activity is shown by both S-carvedilol and R-carvedilol.
Time Frame: Week 8
Population: PK Parameter Population: total of 13 participants, including 3 who gave samples in group F at Week 8 in CRV-IR group; total of 15 participants, including 4 who gave samples at Week 8 in the SK&F-105517-D group)
Measure: Geometric Mean (95% Confidence Interval); unit: nanograms per milliliter (ng/mL)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 3 | 4
nanograms per milliliter (ng/mL)
  S-carvedilol, Cmax | 6.7952 [5.8993 to 7.8272] | 12.8171 [3.6610 to 44.8731]
  S-carvedilol, Cmin | 1.2072 [0.1282 to 11.3641] | 3.3796 [1.8809 to 6.0727]
  R-carvedilol, Cmax | 19.1864 [9.3670 to 39.2994] | 27.1306 [8.9369 to 82.3626]
  R-carvedilol, Cmin | 2.9445 [1.7119 to 5.0647] | 4.2565 [2.3297 to 7.7768]
  SB-203231, Cmax | 3.1665 [2.5819 to 3.8833] | 6.3937 [2.3918 to 17.0913]
  SB-203231, Cmin | 0.4843 [0.2322 to 1.0101] | 1.2386 [0.7761 to 1.9769]

3. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time Zero to 24 Hours (AUC0-24) of S-carvedilol, R-carvedilol, and M4 Active Metabolite (SB-203231) at Week 8
Description: Area under the plasma concentration versus time curve from time zero to 24 hours (AUC0-24) of S-carvedilol, R-carvedilol, and M4 active metabolite (SB-203231) was measured. Participants in each treatment group were divided into 3 groups by pharmacokinetic sampling timing: Groups A, B, and C in the SK&F-105517-D group and Groups D, E, and F in the CRV-IR group. The analysis was performed on log-transformed data. Carvedilol is a racemic mixture. Non-selective β-blocking activity is shown by S-carvedilol, while α1-blocking activity is shown by both S-carvedilol and R-carvedilol.
Time Frame: Week 8
Population: Pharmacokinetic (PK) Parameter Population: all participants who received the study drug at each dose level and provided sufficient PK concentration data and the data for estimation of PK parameters (total of 13 participants, 3 gave samples at Week 8 in CRV-IR group; total of 15 participants, 4 gave samples at Week 8 in the SK&F-105517-D group)
Measure: Geometric Mean (95% Confidence Interval); unit: hours * nanograms per milliliter (ng/mL)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 3 | 4
hours * nanograms per milliliter (ng/mL)
  S-carvedilol | 60.040 [12.856 to 280.396] | 155.109 [63.319 to 379.959]
  R-carvedilol | 170.728 [131.607 to 221.478] | 284.313 [132.307 to 610.954]
  SB-203231 | 28.113 [14.853 to 53.209] | 64.687 [28.012 to 149.382]

4. Secondary Outcome: Time of Maximal Plasma Concentration (Tmax) of S-carvedilol, R-carvedilol, and M4 Active Metabolite (SB-203231) at Week 8
Description: Time of maximal plasma concentration (tmax) of S-carvedilol, R-carvedilol, and M4 active metabolite (SB-203231) was measured. Participants in each treatment group were divided into 3 groups by pharmacokinetic sampling timing: Groups A, B, and C in the SK&F-105517-D group and Groups D, E, and F in the CRV-IR group. Carvedilol is a racemic mixture. Non-selective β-blocking activity is shown by S-carvedilol, while α1-blocking activity is shown by both S-carvedilol and R-carvedilol.
Time Frame: Week 8
Population: PK Parameter Population: total of 13 participants, including 3 in group F who gave samples at Week 8 in the CRV-IR group; total of 15 participants, including 4 in group C who gave samples at Week 8 in the SK&F-105517-D group
Measure: Median (Full Range); unit: hours
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 3 | 4
hours
  S-carvedilol | 1.983 [1.00 to 2.03] | 5.958 [4.00 to 6.08]
  R-carvedilol | 1.983 [1.00 to 2.03] | 5.958 [4.00 to 6.08]
  SB-203231 | 1.983 [1.00 to 2.03] | 5.958 [4.00 to 6.08]

5. Secondary Outcome: Adjusted Mean Change From Baseline in Systolic Blood Pressure at Week 8
Description: Pharmacodynamic (PD) assessment points were 24 hours (h) (from time of first reading to time of last reading), morning (6 am-12 pm), afternoon (12-6 pm), night (6 pm-6 am on following day), waking (8 am-9 pm), sleeping (0-5 am), PDmax (maximal value obtained with each participant during the 0-24 h interval), PDmin (minimal value obtained with each participant during the 0-24 h interval), and PDmax/PDmin. PDmax/PDmim was calculated as the ratio of the PDmax to PDmin, and it showed the degree of change during the 0-24 h interval. The mean was adjusted for Baseline value.
Time Frame: Baseline and Week 8
Population: Pharmacodynamic (PD) Population: all participants measurable at the PD endpoints (18 participants at baseline and 3 participants at Week 8 in CRV-IR group, 19 participants at baseline and 4 participants at Week 8 in SK&F-105517-D group)
Measure: Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 18 | 19
millimeters of mercury (mmHg)
  24 h | -10.84 (4.119) | -1.45 (3.567)
  Morning | -12.34 (4.412) | -4.78 (3.819)
  Afternoon | -10.14 (2.734) | -12.06 (2.361)
  Night | -9.04 (4.786) | 5.17 (4.139)
  Waking | -10.39 (2.857) | -9.99 (2.472)
  Sleeping | -11.85 (3.223) | 13.20 (2.787)
  PDmax | -9.74 (7.772) | -10.19 (6.656)
  PDmin | -6.89 (5.416) | 1.42 (4.685)
  PDmax/PDmin | 0.07 (0.103) | -0.17 (0.088)
Statistical Analysis 1: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = 9.38, 95% CI 2-sided [-5.75 to 24.51], Standard Error of Mean 5.449 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the 24 h assessment
Statistical Analysis 2: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Median Difference (Net) = 7.55, 95% CI 2-sided [-8.68 to 23.79], Standard Error of Mean 5.849 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Morning assessment
Statistical Analysis 3: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -1.92, 95% CI 2-sided [-12.04 to 8.20], Standard Error of Mean 3.645 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Afternoon assessment
Statistical Analysis 4: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = 14.21, 95% CI 2-sided [-3.45 to 31.87], Standard Error of Mean 6.361 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Night assessment
Statistical Analysis 5: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = 0.40, 95% CI 2-sided [-10.12 to 10.92], Standard Error of Mean 3.790 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Waking assessment
Statistical Analysis 6: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = 25.04, 95% CI 2-sided [13.16 to 36.93], Standard Error of Mean 4.281 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Sleeping assessment
Statistical Analysis 7: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -0.45, 95% CI [-29.94 to 29.03], Standard Error of Mean 10.62 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the PDmax assessment
Statistical Analysis 8: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = 8.31, 95% CI 2-sided [-11.67 to 28.28], Standard Error of Mean 7.194 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the PDmin assessment
Statistical Analysis 9: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -0.24, 95% CI 2-sided [-0.63 to 0.15], Standard Error of Mean 0.142 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the PDmax/PDmin assessment

6. Primary Outcome: Mean Change From Baseline in Albumin and Total Protein at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: Safety Population: 22 participants at baseline and 11 participants at Week 8 in the CRV-IR group; 19 participants at baseline and 8 participants at Week 8 in the SK&F-105517-D group. Some participants in each treatment arm withdrew prematurely.
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
grams per liter (g/L)
  Albumin | 0.7 (2.87) | -1.9 (2.90)
  Total Protein | 0.4 (4.27) | -1.6 (4.72)

7. Primary Outcome: Mean Change From Baseline in Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, Creatine Kinase, and Gamma Glutamyl Transferase at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: international units per liter (IU/L)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
international units per liter (IU/L)
  Alkaline Phosphatase | -10.9 (18.45) | -5.0 (21.13)
  Alanine Aminotransferase | -0.2 (6.48) | 3.8 (9.39)
  Aspartate Aminotransferase | 0.8 (3.87) | 1.4 (7.19)
  Creatine Kinase | 34.4 (55.58) | -0.1 (65.54)
  Gamma Glutamyl Transferase | -0.8 (3.68) | 2.4 (10.62)

8. Primary Outcome: Mean Change From Baseline in Amylase at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units per liter (U/L)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
units per liter (U/L) | -10.2 (9.98) | -0.1 (15.66)

9. Primary Outcome: Mean Change From Baseline in Total Bilirubin, Creatinine, and Uric Acid at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: micromoles per liter (umol/L)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
micromoles per liter (umol/L)
  Total Bilirubin | 1.555 (2.3514) | -4.489 (3.8712)
  Creatinine | 5.5451 (14.97638) | -4.5305 (5.85307)
  Uric Acid | 30.8215 (48.16177) | 14.1265 (80.67868)

10. Primary Outcome: Mean Change From Baseline in Calcium, Chloride, Glucose, Potassium, Sodium, and Urea/Blood Urea Nitrogen at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
millimoles per liter (mmol/L)
  Calcium | -0.027218 (0.1364081) | -0.056138 (0.0592680)
  Chloride | 0.2 (1.60) | 2.4 (2.20)
  Glucose | -0.136252 (2.9159783) | -1.956728 (2.8733368)
  Potassium | -0.07 (0.361) | 0.07 (0.474)
  Sodium | 0.5 (2.30) | 1.6 (1.41)
  Urea/Blood Urea Nitrogen | 0.61339 (2.523049) | -0.58013 (1.023316)

11. Primary Outcome: Mean Change From Baseline in Creatine Kinase BB Percentage, Creatine Kinase MB Percentage, and Creatine Kinase MM Percentage at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value. (BB, brain-derived; MB=cardiac muscle-derived; MM=skeletal muscle-derived.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of Total Creatine Kinase
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
percentage of Total Creatine Kinase
  Creatine Kinase BB percentage | -0.2 (0.60) | 0.5 (0.93)
  Creatine Kinase MB percentage | -0.3 (0.65) | -0.1 (0.83)
  Creatine Kinase MM percentage | 1.1 (1.30) | 0.8 (1.75)

12. Primary Outcome: Mean Change From Baseline in Each Type of White Blood Cell (WBC) (Basophils, Eosinophils, Lymphocytes, Monocytes, and Total Neutrophils) at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of each WBC type in WBC count
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
percentage of each WBC type in WBC count
  Basophils | -0.06 (0.403) | -0.06 (0.325)
  Eosinophils | 0.15 (1.547) | 0.76 (1.412)
  Lymphocytes | 0.05 (6.052) | 2.21 (9.174)
  Monocytes | 0.19 (1.358) | 1.28 (1.356)
  Total Neutrophils | -0.41 (7.875) | -4.31 (11.180)

13. Primary Outcome: Mean Change From Baseline in Hemoglobin and Mean Corpuscular Hemoglobin Concentration at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: grams per liter (g/L)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
grams per liter (g/L)
  Hemoglobin | -2.3 (8.05) | -3.9 (8.04)
  Mean Corpuscular Hemoglobin Concentration | 1.3 (4.90) | -1.9 (6.01)

14. Primary Outcome: Mean Change From Baseline in Hematocrit at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: proportion of 1 (SI)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
proportion of 1 (SI) | -0.0085 (0.02306) | -0.0095 (0.02287)

15. Primary Outcome: Mean Change From Baseline in Platelet Count and White Blood Cell Count at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: gibi (2 to the power of 30)/liter (Gi/L)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
gibi (2 to the power of 30)/liter (Gi/L)
  Platelet Count | -6.9 (23.28) | -11.1 (14.54)
  White Blood Cell Count | 0.297 (0.9850) | -0.498 (1.9516)

16. Primary Outcome: Mean Change From Baseline in Red Blood Cell Count at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: tebi (2 to the power of 40)/liter (Ti/L)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
tebi (2 to the power of 40)/liter (Ti/L) | -0.091 (0.2390) | -0.087 (0.2295)

17. Primary Outcome: Mean Change From Baseline in Mean Corpuscular Hemoglobin at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
picograms (pg) | 0.12 (0.515) | -0.21 (0.372)

18. Primary Outcome: Mean Change From Baseline in Mean Corpuscular Volume at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: femtoliters (fL)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
femtoliters (fL) | 0.1 (1.38) | -0.1 (1.96)

19. Primary Outcome: Number of Participants With the Indicated Urinalysis Dipstick Results at Baseline and Week 8
Description: Dipstick test values: Negative (-), Traces (+-), +1, +2, +3. +4. Normal ranges (qualitative): protein, - or +-; glucose, - or +-; occult blood, -; ketones, -.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
participants
  Urine Glucose, Negative, Baseline, n=22, 19 | 20 | 19
  Urine Glucose, Traces, Baseline, n=22, 19 | 1 | 0
  Urine Glucose, 1+, Baseline, n=22, 19 | 0 | 0
  Urine Glucose, 2+, Baseline, n=22, 19 | 0 | 0
  Urine Glucose, 3+, Baseline, n=22, 19 | 1 | 0
  Urine Glucose, 4+, Baseline, n=22, 19 | 0 | 0
  Urine Ketones, Negative, Baseline, n=22, 19 | 22 | 19
  Urine Ketones, Traces, Baseline, n=22, 19 | 0 | 0
  Urine Ketones, 1+, Baseline, n=22, 19 | 0 | 0
  Urine Ketones, 2+, Baseline, n=22, 19 | 0 | 0
  Urine Ketones, 3+, Baseline, n=22, 19 | 0 | 0
  Urine Ketones, 4+, Baseline, n=22, 19 | 0 | 0
  Urine Occult Blood, Negative, Baseline, n=22, 19 | 18 | 16
  Urine Occult Blood, Traces, Baseline, n=22, 19 | 1 | 1
  Urine Occult Blood, 1+, Baseline, n=22, 19 | 2 | 1
  Urine Occult Blood, 2+, Baseline, n=22, 19 | 1 | 1
  Urine Occult Blood, 3+, Baseline, n=22, 19 | 0 | 0
  Urine Occult Blood, 4+, Baseline, n=22, 19 | 0 | 0
  Urine Protein, Negative, Baseline, n=22, 19 | 21 | 18
  Urine Protein, Traces, Baseline, n=22, 19 | 0 | 0
  Urine Protein, 1+, Baseline, n=22, 19 | 0 | 1
  Urine Protein, 2+, Baseline, n=22, 19 | 1 | 0
  Urine Protein, 3+, Baseline, n=22, 19 | 0 | 0
  Urine Protein, 4+, Baseline, n=22, 19 | 0 | 0
  Urine Glucose, Negative, Week 8, n=11, 8 | 11 | 8
  Urine Glucose, Traces, Week 8, n=11, 8 | 0 | 0
  Urine Glucose, 1+, Week 8, n=11, 8 | 0 | 0
  Urine Glucose, 2+, Week 8, n=11, 8 | 0 | 0
  Urine Glucose, 3+, Week 8, n=11, 8 | 0 | 0
  Urine Glucose, 4+, Week 8, n=11, 8 | 0 | 0
  Urine Ketones, Negative, Week 8, n=11, 8 | 11 | 8
  Urine Ketones, Traces, Week 8, n=11, 8 | 0 | 0
  Urine Ketones, 1+, Week 8, n=11, 8 | 0 | 0
  Urine Ketones, 2+, Week 8, n=11, 8 | 0 | 0
  Urine Ketones, 3+, Week 8, n=11, 8 | 0 | 0
  Urine Ketones, 4+, Week 8, n=11, 8 | 0 | 0
  Urine Occult Blood, Negative, Week 8, n=11, 8 | 11 | 8
  Urine Occult Blood, Traces, Week 8, n=11, 8 | 0 | 0
  Urine Occult Blood, 1+, Week 8, n=11, 8 | 0 | 0
  Urine Occult Blood, 2+, Week 8, n=11, 8 | 0 | 0
  Urine Occult Blood, 3+, Week 8, n=11, 8 | 0 | 0
  Urine Occult Blood, 4+, Week 8, n=11, 8 | 0 | 0
  Urine Protein, Negative, Week 8, n=11, 8 | 10 | 8
  Urine Protein, Traces, Week 8, n=11, 8 | 1 | 0
  Urine Protein 1+, Week 8, n=11, 8 | 0 | 0
  Urine Protein, 2+, Week 8, n=11, 8 | 0 | 0
  Urine Protein, 3+, Week 8, n=11, 8 | 0 | 0
  Urine Protein, 4+, Week 8, n=11, 8 | 0 | 0

20. Primary Outcome: Mean Change From Baseline in Systolic Blood Pressure and Diastolic Blood Pressure at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
millimeters of mercury (mmHg)
  Systolic blood pressure | -5.7 (20.68) | 10.0 (15.28)
  Diastolic blood pressure | 0.6 (11.69) | 2.8 (5.68)

21. Primary Outcome: Mean Change From Baseline in Heart Rate at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
beats per minute | -10.4 (10.54) | -10.6 (18.87)

22. Primary Outcome: Mean Change From Baseline in Weight at Week 8
Description: Mean change from baseline was calculated as the Week 8 value minus the Baseline value.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
kilograms (kg) | 0.29 (1.490) | -0.11 (2.303)

23. Primary Outcome: Number of Participants With the Indicated Electrocardiogram Findings at Baseline and Week 8
Description: There are 3 categories for electrocardiogram (ECG) findings: normal; abnormal, not clinically significant; and abnormal, clinically significant. Each of the findings was classified by the investigator according to whether it was normal. Abnormal ECGs were further classified according to whether they were felt to be clinically significant in the medical and scientific judgment of the investigator.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
participants
  Normal, Baseline (BL), n=22, 19 | 2 | 1
  Abnormal-Not clinically significant, BL, n=22, 19 | 12 | 9
  Abnormal-Clinically significant, BL, n=22, 19 | 8 | 9
  Normal, Week (W) 8, n=11, 8 | 2 | 1
  Abnormal-Not clinically significant, W8, n=11, 8 | 5 | 1
  Abnormal-Clinically significant, W8, n=11, 8 | 4 | 6

24. Primary Outcome: Cardiothoracic Ratio at Baseline and Week 8
Description: Cardiothoracic ratio is a marker of the degree of heart enlargement and was measured by chest X-ray. It is shown as the ratio of the transverse diameter of the heart to the transverse diameter of the thorax, and is measured as a percentage.
Time Frame: Baseline and Week 8
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 22 | 19
percentage
  Baseline, n=22, 19 | 53.70 (4.536) | 53.58 (8.098)
  Week 8, n=11, 8 | 50.91 (4.309) | 52.35 (7.545)

25. Secondary Outcome: Adjusted Mean Change From Baseline in Diastolic Blood Pressure at Week 8
Description: as for outcome 5
Time Frame: Baseline and Week 8
Population: as for outcome 5
Measure: Mean (Standard Error); unit: millimeters of mercury (mmHg)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 18 | 19
millimeters of mercury (mmHg)
  24 h | -7.10 (3.387) | -4.89 (2.852)
  Morning | -7.68 (4.449) | -8.24 (3.766)
  Afternoon | -5.32 (2.760) | -10.25 (2.336)
  Night | -9.01 (4.190) | 0.73 (3.506)
  Waking | -5.11 (2.902) | -8.56 (2.458)
  Sleeping | -12.68 (1.197) | 5.38 (1.011)
  PDmax | -10.45 (6.702) | -17.91 (5.796)
  PDmin | -1.34 (3.852) | -0.24 (3.291)
  PDmax/PDmin | -0.24 (0.111) | -0.36 (0.094)
Statistical Analysis 1: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = 2.21, 95% CI 2-sided [-11.20 to 15.63], Standard Error of Mean 4.833 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the 24 h assessment
Statistical Analysis 2: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -0.56, 95% CI 2-sided [-17.95 to 16.84], Standard Error of Mean 6.265 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Morning assessment
Statistical Analysis 3: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -4.93, 95% CI 2-sided [-15.71 to 5.86], Standard Error of Mean 3.885 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Afternoon assessment
Statistical Analysis 4: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = 9.74, 95% CI 2-sided [-7.11 to 26.59], Standard Error of Mean 6.070 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Night assessment
Statistical Analysis 5: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -3.45, 95% CI 2-sided [-14.78 to 7.88], Standard Error of Mean 4.080 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Waking assessment
Statistical Analysis 6: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = 18.06, 95% CI 2-sided [13.36 to 22.76], Standard Error of Mean 1.694 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Sleeping assessment
Statistical Analysis 7: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -7.46, 95% CI 2-sided [-32.17 to 17.26], Standard Error of Mean 8.902 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the PDmax assessment
Statistical Analysis 8: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = 1.10, 95% CI 2-sided [-13.61 to 15.80], Standard Error of Mean 5.297 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the PDmin assessment
Statistical Analysis 9: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -0.12, 95% CI 2-sided [-0.54 to 0.30], Standard Error of Mean 0.152 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the PDmax/PDmin assessment

26. Secondary Outcome: Adjusted Mean Change From Baseline in Mean Heart Rate at Week 8
Description: as for outcome 5
Time Frame: Baseline and Week 8
Population: PD Population: all participants measurable at the PD endpoints (18 participants at baseline and 3 participants at Week 8 in CRV-IR group, 19 participants at baseline and 4 participants at Week 8 in SK&F-105517-D group)
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 18 | 19
beats per minute
  24 h | -11.38 (2.385) | -15.37 (2.058)
  Morning | -9.59 (2.225) | -14.87 (1.923)
  Afternoon | -13.96 (2.345) | -15.93 (2.006)
  Night | -11.12 (2.760) | -15.26 (2.387)
  Waking | -12.53 (2.250) | -15.53 (1.933)
  Sleeping | -11.16 (3.536) | -14.28 (3.060)
  PDmax | -13.43 (2.758) | -23.43 (2.366)
  PDmin | -2.04 (3.830) | -3.47 (3.276)
  PDmax/PDmin | -0.93 (0.095) | -1.27 (0.080)
Statistical Analysis 1: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -3.99, 95% CI 2-sided [-12.84 to 4.86], Standard Error of Mean 3.187 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the 24 h assessment
Statistical Analysis 2: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -5.27, 95% CI 2-sided [-13.50 to 2.95], Standard Error of Mean 2.962 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Morning assessment
Statistical Analysis 3: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -1.98, 95% CI 2-sided [-10.89 to 6.94], Standard Error of Mean 3.209 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Afternoon assessment
Statistical Analysis 4: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -4.14, 95% CI 2-sided [-14.32 to 6.03], Standard Error of Mean 3.665 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Night assessment
Statistical Analysis 5: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -2.99, 95% CI 2-sided [-11.45 to 5.47], Standard Error of Mean 3.047 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Waking assessment
Statistical Analysis 6: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -3.11, 95% CI 2-sided [-16.12 to 9.89], Standard Error of Mean 4.686 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the Sleeping assessment
Statistical Analysis 7: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -10.00, 95% CI 2-sided [-20.41 to 0.41], Standard Error of Mean 3.749 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the PDmax assessment
Statistical Analysis 8: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -1.42, 95% CI 2-sided [-16.00 to 13.15], Standard Error of Mean 5.249 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the PDmin assessment
Statistical Analysis 9: Comparison: CRV-IR vs SK&F-105517-D; Test type: Superiority or Other; Mean Difference (Net) = -0.34, 95% CI 2-sided [-0.71 to 0.03], Standard Error of Mean 0.133 — The mean treatment difference is calculated as SK&F-105517-D minus CRV-IR for the PDmax/PDmin assessment

27. Secondary Outcome: Number of Participants With the Indicated Change From Baseline New York Heart Association (NYHA) Functional Class at Week 8
Description: The NYHA classification assesses the severity of symptoms of heart failure as judged by the investigator and is comprised of. 4 classes: I, no resulting limitations on physical activity (PA); II, slight limitations on PA; III, marked limitations on PA; IV, inability to carry out any PA without discomfort. The number of participants with any change from Baseline in the NYHA Functional Class at Week 8 was calculated. Improved=class at the visit is decreased compared to baseline class, Unchanged=class at the visit is stable, Worsened=class at the visit is increased compared to baseline class.
Time Frame: Baseline and Week 8
Population: Efficacy Population: all participants measurable at the efficacy endpoints (20 participants at baseline and 11 participants at Week 8 in the CRV-IR group; 19 participants at baseline and 8 participants at Week 8 in the SK&F-105517-D group. Some participants in each treatment arm withdrew prematurely.
Measure: Number; unit: participants
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 20 | 19
participants
  Improved | 0 | 1
  Unchanged | 11 | 7
  Worse | 0 | 0

28. Secondary Outcome: Mean Plasma Brain Natriuretic Peptide Concentration at Baseline and Week 8
Description: Brain natriuretic peptide is a surrogate marker of the severity of heart failure and was measured by a central laboratory.
Time Frame: Baseline and Week 8
Population: Efficacy Population: all participants measurable at the efficacy endpoints (20 participants at baseline and 11 participants at Week 8 in the CRV-IR group; 19 participants at baseline and 8 participants at Week 8 in the SK&F-105517-D group). Some participants in each treatment arm withdrew prematurely.
Measure: Mean (Standard Deviation); unit: ng/L (nanogram per Liter)
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 20 | 19
ng/L (nanogram per Liter)
  Baseline, n=20, 19 | 108.93 (112.192) | 226.46 (339.640)
  Week 8, n=11, 8 | 64.88 (62.020) | 111.93 (84.298)

29. Secondary Outcome: Echocardiogram Results: Left Ventricular Ejection Fraction at Baseline and Week 8
Description: Left ventricular ejection fraction (LVEF) is a marker of left ventricular systolic function and was measured by echocardiogram. It is shown as the ratio of left ventricular stroke volume (LVSV) to left ventricular end-diastolic volume (LVEDV), and is measured as a percentage.
Time Frame: Baseline and Week 8
Population: as for outcome 28
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | CRV-IR | SK&F-105517-D
Number analyzed (Participants) | 20 | 19
percentage
  Baseline, n=20, 19 | 34.0 (8.43) | 32.2 (10.09)
  Week 8, n=11, 8 | 42.0 (13.36) | 37.6 (10.14)

ADVERSE EVENTS:
Time Frame: Treatment Period from Week 0 (Baseline) to Week 8 and 1-week Follow-up Period (Week 9) for CRV-IR; Treatment Period from Week 0 (Baseline) to Week 14 and 1-week Follow-up Period (Week 15) for SK&F-105517-D.
Arm/Group | CRV-IR | SK&F-105517-D
Serious Adverse Events (participants affected / at risk) | 1/22 | 3/19
Other Adverse Events (participants affected / at risk) | 11/22 | 15/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CRV-IR (N=22) | SK&F-105517-D (N=19)
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CRV-IR (N=22) | SK&F-105517-D (N=19)
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Nasopharyngitis (Infections and infestations) | 2 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 2
Dizziness (Nervous system disorders) | 1 | 2
Blood uric acid increased (Investigations) | 1 | 1
Brain natriuretic peptide increased (Investigations) | 1 | 1
Bronchitis (Infections and infestations) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood calcium decreased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Nodal rhythm (Cardiac disorders) | 0 | 1
Platelet count decreased (Investigations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.